CLINICAL TRIAL: NCT06040515
Title: Probiotic EcN in Symptomatic Patients After an Episode of Acute Colonic Diverticulitis: a Prospective Multicentre Observational Study.
Brief Title: Probiotic After Acute Colonic Diverticulitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmo Spaziani (Other)
Responsible Party: Sponsor-Investigator, Erasmo Spaziani, MD, PhD, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Other Study IDs: EcN2023
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Diverticulitis, Colonic; Therapy
MeSH Terms: conditions — Diverticulitis, Colonic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Symptomatic patients after acute diverticulitis: Patients aged ≥18 with persistent symptoms at least three months after a radiologic and/or endoscopic documented acute diverticulitis or after six months of surgery for complicated acute diverticulitis.
  Therapy with Escherichia coli Nissle 1917 (EcN®) will be prescribed for a global duration of six months with the following assumption schedule: 2 capsules b.i.d. during 4 weeks, followed by 1 capsule o.i.d during 20 days each month for 5 months.
  Interventions: Drug: Probiotic Formula
- Diverticulosis: Patients with asymptomatic diverticulosis. No therapy will be administered. Microbiota assessment will be performed.
- Asymptomatic patients after acute uncomplicated diverticulitis: Asymptomatic patients assessed three months after an episode of acute uncomplicated diverticulitis. No therapy will be administered. Microbiota assessment will be performed.
- Asymptomatic patients after acute complicated diverticulitis: Asymptomatic patients assessed six months after an episode of acute complicated diverticulitis submitted to surgery with resection and without stoma . No therapy will be administered. Microbiota assessment will be performed.

INTERVENTIONS:
Drug: Probiotic Formula — Capsule with 25 billion live strains of Escherichia coli Nissle 1917
  Other Names: Escherichia coli Nissle 1917
  Groups: Symptomatic patients after acute diverticulitis

SUMMARY:
The goal of this observational study is to assess the efficacy and safety of the probiotic Escherichia coli Nissle 1917 (EcN®, Ca.Di.Group S.p.A) in the treatment of symptomatic patients after an episode of both complicated and uncomplicated acute colonic diverticulitis.

The main question it aims to answer are:

* Is the studied probiotic able to significantly reduce symptoms, assessed by means of a validated and dedicated score?
* Is there any difference in microbiota among the study group at baseline and a selected cohort of patients subdivided in subjects with diverticulosis and asymptomatic subjects after an episode of acute uncomplicated diverticulitis or an episode of complicated diverticulitis submitted to surgery with colonic resection without stoma?
* Is there any difference in microbiota in the study group at baseline and after 3 and 6 months of treatment with the probiotic?
* Is there any correlation between microbiota modification and symptoms during follow-up?
* Is there any impact on fecal calprotectin values before and during probiotic therapy?
* Is there any modification of evacuation before and during follow-up?
* Is probiotic able to prevent recurrent episodes of acute diverticulitis during follow-up?
* The safety of the probiotic will be assessed during the follow-up. The study group will be assessed at baseline and during follow-up with a dedicated clinical score and Bristol stool scale. Microbiota and fecal calprotectin values will be also assessed at baseline and during follow-up. Microbiota at baseline will be also evaluated for comparison in the three selected groups with diverticulosis and both asymptomatic and symptomatic after an episode of acute diverticulitis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients three months after an episode of uncomplicated acute colonic diverticulitis;
* Symptomatic patients six months after an episode of complicated acute colonic diverticulitis; submitted to .surgical colonic resection without stoma;
* Patients with diverticulosis;
* Asymptomatic patients three months after an episode of uncomplicated acute colonic diverticulitis;
* Asymptomatic patients six months after an episode of complicated acute colonic diverticulitis; submitted to surgical colonic resection without stoma.

Exclusion Criteria:

* Ongoing acute diverticulitis at radiologic assessment
* Antibiotic therapy, both systemic and topic, and/or probiotics and/or mesalazine within four weeks before enrolment;
* Lactulose-lactitol use within four weeks before enrolment;
* Presence of chronic inflammatory bowel diseases;
* Presence of Segmental Colitis Associated with Diverticulitis (SCAD);
* Presence of ischemic colitis;
* Severe chronic liver (Child-Pugh C) and/or pancreatic and/or renal diseases;
* Patients with severe renal failure;
* Presence of suspected/actual pregnancy;
* Presence of recent/ongoing neoplasia, under oncological treatment within 6 months before enrolment;
* Presence of COVID-19 infection;
* Patients unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include the above specified study groups.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Median symptomatic score reduction after therapy with Escherichia coli Nissle 1917 | Six-months follow-up
  Median symptomatic score assessed at baseline and during follow-up

SECONDARY OUTCOMES:
Microbiota qualitative composition | Baseline
  Composition of microbiota will be assessed in all the study groups with a dedicated kit for collection.
Microbiota qualitative composition modification | Baseline and during 6-month follow-up.
  Composition of microbiota will be assessed in symptomatic study groups with a dedicated kit for collection.
Microbiota qualitative composition and median symptomatic score correlation | Baseline and during 6-month follow-up.
  Correlation between the median symptomatic score and qualitative composition of microbiota modification after therapy.
Concentration of fecal calprotectin | Baseline and during 6-month follow-up.
  Assessment of fecal calprotectin concentration in the symptomatic study group.
Bristol stool scale modification | Baseline and during 6-month follow-up.
  Assessment of median Bristol stool scale in the symptomatic study group.
Prevention of recurrent acute diverticulitis | Six-month follow-up.
  Number off patients with recurrent acute diverticulitis.
Safety | Six-month follow-up.
  Number of patients with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Elisei, MD, Principal Investigator — • UOC di Gastroenterologia, Azienda Ospedaliera "S. Camillo-Forlanini", Roma
Locations (12):
- Italy (12):
  - UOC di Gastroenterologia ed Endoscopia Digestiva, Ospedale "Pugliese-Ciaccio, Catanzaro, Calabria
  - UOSVD di Endoscopia Digestiva, Ospedale "S. Maria Goretti", Latina, Lazio
  - UOC di Gastroenterologia, Azienda Ospedaliera "S. Camillo-Forlanini", Rome, Lazio
  - UOSVD di Gastroenterologia ed Endoscopia Digestiva, Ospedale "Umberto I", Rome, Lazio
  - UOC di Medicina Interna e Gastroenterologia, Ospedale "Cristo Re", Rome, Lazio
  - UOC Chirurgia Generale, Ospedale "P. Colombo", Velletri, Lazio
  - UOC di Gastroenterologia, Ospedale "Belcolle",, Viterbo, Lazio
  - • UOC di Gastroenterologia ed Endoscopia Digestiva, Ospedale Universitario "San Raffaele", Milan, Lombardy
  - UOC di Gastroenterologia Azienda Ospedaliero-Universitaria di Padova, Padova, Lombardy
  - UOC di Gastroenterologia, Ospedale "Guglielmo da Saliceto", Piacenza, Lombardy
  - UOC di Gastroenterologia, Ospedale "S. Salvatore",, Pesaro, The Marches
  - Gastroenterology Service , ASL BAT,, Andria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kvasnovsky CL, Adams K, Papagrigoriadis S. Diverticular disease as a chronic gastrointestinal condition: experience from a specialist clinic. Eur J Gastroenterol Hepatol. 2015 Apr;27(4):442-8. doi: 10.1097/MEG.0000000000000304. PMID 25874519
- [Result] Mj O, Turner GA, A S, Frizelle FA, R P. Distinct changes in the colonic microbiome associated with acute diverticulitis. Colorectal Dis. 2022 Dec;24(12):1591-1601. doi: 10.1111/codi.16271. Epub 2022 Aug 11. PMID 35950499
- [Result] Tursi A, Papa V, Lopetuso LR, Settanni CR, Gasbarrini A, Papa A. Microbiota Composition in Diverticular Disease: Implications for Therapy. Int J Mol Sci. 2022 Nov 26;23(23):14799. doi: 10.3390/ijms232314799. PMID 36499127
- [Result] Teng G, Liu Z, Liu Y, Wu T, Dai Y, Wang H, Wang W. Probiotic Escherichia coli Nissle 1917 Expressing Elafin Protects Against Inflammation and Restores the Gut Microbiota. Front Microbiol. 2022 May 6;13:819336. doi: 10.3389/fmicb.2022.819336. eCollection 2022. PMID 35602072
- [Result] Lahat A, Fidder HH, Ben-Horin S. Development and validation of a diverticular clinical score for symptomatic uncomplicated diverticular disease after acute diverticulitis in a prospective patient cohort. Therap Adv Gastroenterol. 2020 May 8;13:1756284820913210. doi: 10.1177/1756284820913210. eCollection 2020. PMID 32523619